CLINICAL TRIAL: NCT00315653
Title: Evaluation of the Survivin Urine mRNA Assay to Estimate Risk of Bladder Cancer Found on Cystoscopy
Brief Title: Survivin Urine mRNA Assay Risk of Bladder Cancer Study
Status: Completed | Type: Observational
Sponsor: Fujirebio Diagnostics, Inc. (Industry)
Responsible Party: Jeff Allard, PhD, Fujirebio Diagnostics, inc
Other Study IDs: FDI-01 Sure Study
Record Dates: First submitted 2006-04-18; First posted 2006-04-19 (Estimated); Last update posted 2008-03-14 (Estimated); Status verified 2008-03

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Cancer of Bladder; Bladder Tumors; Cancer of the Bladder; Neoplasms, Bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this clinical trial is to evaluate the ability of urinary Survivin mRNA measurement to estimate the risk of bladder cancer at the time of cystoscopy in subjects with no prior history of bladder cancer presenting with microscopic or macroscopic hematuria.

DETAILED DESCRIPTION:
Bladder cancer is the fourth most common cancer in men and ninth most common cancer in women, accounting for more than 60,000 new cases and ~12,000 deaths in North America in 2004. Cystoscopy and urinary cytology is the standard of care for detection of bladder cancer, but cystoscopy is expensive and invasive, while cytology has low sensitivity. New, noninvasive, diagnostic tools for bladder cancer detection have been developed, but their application in clinical practice has been limited due to low sensitivity and specificity of the assays. Survivin, an anti-apoptotic protein, is capable of regulating both cell proliferation and apoptotic cell death, and is over-expressed in most human cancers but not in normal adult tissues. The purpose of this clinical trial is to evaluate the ability of urinary Survivin mRNA measurement to estimate the risk of bladder cancer at the time of cystoscopy in subjects with no prior history of bladder cancer presenting with microscopic or macroscopic hematuria.

This study is designed to be a prospective, multicenter, double blind, clinical study in subjects >50 years old with no prior history of bladder cancer and confirmed hematuria (microscopic and/or macroscopic) presenting to a urologist.

The primary objective of the study is to estimate the risk of bladder cancer at the time of cystoscopy in subjects >50 years old with no prior history of bladder cancer and confirmed hematuria using urinary Survivin mRNA levels.

The secondary objective of the study is for comparison of a multivariate predictive algorithm using urinary Survivin mRNA levels and subject risk factors, such as age, sex, race, and smoking history, for estimation of the risk of bladder cancer at the time of cystoscopy in subjects >50 years old with no prior history of bladder cancer and confirmed hematuria to the use of urinary Survivin mRNA levels alone.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign Informed Consent;
* Age >50 years old;
* Males or females;
* Subjects must have confirmed micro-hematuria, defined as any positive urine reagent strip test for blood (i.e. finding of "Trace" or higher amounts of blood) and/or >3 RBC per high power field on microscopic examination, or macro-hematuria, defined as visible blood in the urine sample;
* All subjects must be scheduled to undergo a cystoscopy evaluation;
* All subjects must have upper tract imaging performed within +/- 4 weeks of the cystoscopic evaluation.

Exclusion Criteria:

* Previous history of bladder cancer;
* Previous history of other cancers except for non-melanoma skin cancer;
* Prior pelvic radiation;
* Active urinary or vaginal infection;
* Any evidence of vaginal or rectal bleeding;
* Currently receiving chemotherapies such as cyclophosphamide or methotrexate;
* Unable to provide informed consent or a high risk that the subject may not comply with the protocol requirements.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects scheduled to undergo cystoscopy
Enrollment: 600
Dates: Start 2005-09; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J Allard, PhD, Study Director — Fujirebio Diagnostics, Inc.; Jose G Moreno, MD, Principal Investigator — Tri County Urologic Associates, PC
Locations (1):
- Fujirebio Diagnostics, Inc, Malvern, Pennsylvania, United States